CLINICAL TRIAL: NCT07153640
Title: EFFECT OF WIM HOF BREATHING EXERCISE ON VENTILATORY FUNCTIONS IN SMOKERS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Eman Kadry Abd Elghany Elnaqeeb, Assistant lectuer, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005934
Record Dates: First submitted 2025-08-16; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-04

CONDITIONS: Smoking Electronic Cigarettes (Vaping), With Moderate and High Dependence for Nicotine
Keywords: WIM HOF BREATHING EXERCISE
MeSH Terms: conditions — Vaping | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind Controlled Clinical Trial (RCT) in which the selected subject will be divided randomly blinded into two groups (21 subjects for study group and 21 subjects for control group). In the study group, subjects in this group will receive Wim Hof Breathing Exercise every day in the morning or at least three hours postprandial and aerobic exercise (5 days/week) for four weeks. Subjects in the control group will receive only aerobic exercise (5 days/week) for four weeks.
  Both groups will be evaluated at baseline and after the end of the treatment program.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomized, Double-blind Controlled Clinical Trial (RCT) in which the selected subject will be divided randomly blinded into two groups (21 subjects for study group and 21 subjects for control group). In the study group, subjects in this group will receive Wim Hof Breathing Exercise every day in the morning or at least three hours postprandial and aerobic exercise (5 days/week) for four weeks. Subjects in the control group will receive only aerobic exercise (5 days/week) for four weeks.
  Both groups will be evaluated at baseline and after the end of the treatment program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wim Hof Breathing Exercise group (Experimental): In the study group, subjects in this group will receive Wim Hof Breathing Exercise every day in the morning or at least three hours postprandial and aerobic exercise (5 days/week) for four weeks.
  Interventions: Other: 1 ) Wim Hof Breathing Exercise; Other: 2) Aerobic exercises
- control group (Active Comparator): Subjects in the control group will receive only aerobic exercise (5 days/week) for four weeks.
  Interventions: Other: 2) Aerobic exercises

INTERVENTIONS:
Other: 1 ) Wim Hof Breathing Exercise — 1. Subjects will be asked to breathe deeply for an average of 20-30 breaths then exhale, (deep rapid inhalations and relaxed expirations)
  2. Hold their breath in an unforced manner for one minute or longer until they feel the urge to breathe (retention phase).
     (For safety, they were instructed not to hold their breath longer than 3.5 min).
  3. Take deep inhalation breath and hold again for 15 seconds (recovery breath).
  4. This procedure was repeated a total of three times.
  5. After the last cycle, subjects were instructed to return to their natural rhythm of breathing and remain lying down without moving to relax for five minutes.
  6. Done every day in the morning or at least three hours postprandial for four weeks.
  (Marko et al., 2022)
  Arms: Wim Hof Breathing Exercise group
Other: 2) Aerobic exercises — Aerobic exercises were performed by walking on the treadmill for 30 minutes a day (5 days/week) and at least 150 minutes per week of moderate-intensity aerobic activity at 60-75% of the maximum heart rate (HR) for four weeks. Maximum heart rate is taken from 220 - to age. Both the warm-up and cool-down were performed for five minutes. Each session concluded with stretching the calf, hamstring, quadriceps, gluteus, back, neck, and shoulder muscles (Acar et al., 2024; Shandu et al., 2023a)

SUMMARY:
Cigarette smoking is the most common form of tobacco use worldwide, but other tobacco products, such as e-cigarettes, cigars, cigarillos, roll-your-own, pipes, and various smokeless tobacco products are also damaging. Most harmful chemicals in cigarette smoke target metals or carbonyls generated by the thermal decomposition of carrier liquids such as propylene glycol, which is one of the main ingredients in the liquid used in electronic cigarettes, where it serves as both the carrier for nicotine and cannabinoids and the means of producing vapor which resemble smoke. This new tobacco product was made of milder sorts of tobacco, the smoke could be inhaled, and it was more damaging.

DETAILED DESCRIPTION:
Smoking primarily causes diseases of the respiratory system, cancer, and the cardiovascular system. E-cigarettes are battery-powered devices that heat a liquid, usually containing nicotine and flavorings, to generate an aerosol for inhalation. In 2014, there were already more than 450 different e-cigarettes with now different generations and more than 8000 different liquids.

The increasing prevalence of smoking among college students presents a significant public health and educational problem, particularly in developing countries where smoking prevention measures are not Strictly enforced .

A healthy lifestyle can reduce the risk of disease. One of the unhealthy lifestyle patterns is consuming cigarettes. Smoking can also reduce the affinity of oxygen for hemoglobin so that it can affect oxygen saturation levels in the blood. Cigarette smoke that enters the body through the lungs contains carbon monoxide and nicotine enters the blood, and then flows throughout the body, and this has an impact on the muscles becoming deprived of oxygen intake, which causes muscle work to be hampered so that the work of the heart will also be hindered because of blockage of blood vessels. It makes the heart pump harder, decreasing the heart's work power.

Wim Hof breathing exercise is part of a structured regimen, called the Wim Hof Method (WHM), which consists of three pillars (breathing, cold exposure, and mindset training). The WHM breathing exercise consists of three or more rounds, each comprising three phases; Hyperventilation, Breath retention, and Recovery breath. The use of Wim Hof breathing method is one of the effective breathing techniques, that increase the level of oxygenation and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* • The age of the subjects ranged from 18-29 years old.

  * The males are participated.
  * Any subjects smoking electronic cigarettes (vaping).
  * Subjects with body mass index between 18.5 - 29.9 Kg/m2.
  * Penn State Electronic Cigarette Dependence Index (moderate and high dependent) (Appendix 1) (Maraqa et al., 2024).

Exclusion Criteria:

* • History of syncope (fainting).

  * High blood pressure (>140/100 mm Hg) (Shandu et al., 2023a).
  * Any type of heart disease.
  * Seizures or Epilepsy.
  * Recent surgery.
  * Metabolic disorders.
  * Subjects with body mass index more than 35 Kg/m2.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
1) Ventilatory Functions | four weeks
  for measuring FVC (forced vital capacity), FEV1(forced expiratory volume in first second), FEV1/FVC (forced expiratory volume in first second /forced vital capacity ratio) and PEF (peak expiratory flow).

SECONDARY OUTCOMES:
1) Functional Capacity | four weeks
  The 6-minute walk distance (6MWD) test for measuring functional capacity. Measured distance by meter.
2) Oxygen saturation | four weeks
  Pulse oximetry provides a noninvasive approximation of the amount of oxygen in arterial blood.
3) Hand grip strength | four weeks
  The gold standard for measuring grip strength is Hydraulic Hand Dynamometer.
4) Smoking Craving | four weeks
  The 10-item Questionnaire on Smoking Urges (QSU-Brief) is a self-report measure designed to assess urges and cravings to smoke, with higher scores indicating stronger urges.
5) Academic Performance | four weeks
  The Academic Performance Scale (APS) is a questionnaire designed to assess academic performance among students based on student self-reports.

CONTACTS AND LOCATIONS:
Overall Officials: EMAN KADRY ELNAQEEB, Master degree, Principal Investigator — October 6 University
Locations (1):
- 6 October, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No